CLINICAL TRIAL: NCT01598194
Title: Prospective Comparison of a Novel 22-gauge Core Biopsy Needle With Reverse Bevel Design to a Standard Endoscopic Ultrasound (EUS) Guided Fine Needle Aspiration (FNA) Needle for Diagnosis of Solid Pancreatic Mass Lesions
Brief Title: Comparison of a Novel 22-gauge Core Biopsy Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-0907
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Solid Pancreatic Mass Lesions; Malignant Neoplasm of Pancreas
Keywords: solid pancreatic mass lesions; 22-gauge core biopsy needle; reverse bevel design; endoscopic ultrasound; EUS; guided; fine needle aspiration; FNA
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Novel 22-gauge Core Biopsy Needle Standard Biopsy Needle (Experimental): The 22-gauge core biopsy needle with reverse bevel design (EchoTip® Procore™) will be compared prospectively to the standard straight hollow-core 22-gauge or 25-gauge FNA needle already used in our clinical practice for the diagnosis of solid pancreatic lesions.
  Interventions: Device: Novel 22-gauge Core Biopsy Needle + Standard Biopsy Needle

INTERVENTIONS:
Device: Novel 22-gauge Core Biopsy Needle + Standard Biopsy Needle — Two passes performed with the standard 22-gauge or 25-gauge straight hollow core needle and two passes will be performed using the 22-gauge EchoTip® Procore™ needle. All passes will be taken from a single lesion and from the same endoscopic location.

SUMMARY:
The goal of this clinical research study is to compare the performance of a newly available needle with reverse bevel design (called the EchoTip® Procore™ needle) with standard needles to see which needle gives better diagnostic information for pancreatic lesions.

DETAILED DESCRIPTION:
An endoscopic ultrasound-guided needle biopsy or FNA is a special endoscopic procedure used to sample lesions within or next to the digestive tract, including the pancreas. The needle is used to collect material for diagnosis. A special lighted, flexible tube called an endoscope is inserted through the mouth, into the stomach and small intestine. The endoscope also has an ultrasound probe at its tip which can be used to see the pancreas, which is located behind the stomach. The doctor will then use the ultrasound to guide the needle biopsy or FNA.

In this procedure, an average of 4 needle passes (needle sticks) is needed to collect enough tissue for diagnosis. However, the number of passes can be higher or lower, depending on the individual lesion and success of the needle passes.

If participant agrees to take part in this study, 2 different needles (the standard straight hollow-core needle and the new EchoTip® Procore™ needle) will be used to sample the pancreas lesion. Two (2) passes will be performed with each needle type and compared. If additional passes are needed for diagnosis, they will not be included in this study. After the first set of needle passes, the doctor may decide that more passes are needed.

Final test results will be taken from the diagnostic results from each needle pass. The results from both types of the needle will be included in the participant's medical record.

This is an investigational study. All needles used in this study are FDA approved and commercially available. Comparing the needles is investigational.

Up to 60 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 years and older.
2. All patients referred for EUS FNA of endoscopically accessible solid pancreatic lesions.

Exclusion Criteria:

1. Unable to obtain informed consent.
2. Unable to tolerate the procedure.
3. Women with known pregnancy at time.
4. Patient age less than 18 years of age.
5. Bleeding diathesis
6. Cystic pancreatic lesions
7. Lesion not accessible by EUS guided FNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Weston, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Weston BR, Ross WA, Bhutani MS, Lee JH, Pande M, Sholl AB, Krishnamurthy S. Prospective randomized comparison of a 22G core needle using standard versus capillary suction for EUS-guided sampling of solid pancreatic masses. Endosc Int Open. 2017 Jun;5(6):E505-E512. doi: 10.1055/s-0043-105492. Epub 2017 Jun 7. PMID 28596983
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 consecutive participants referred for diagnostic EUS-FNA of suspected solid pancreatic mass on CT imaging, recruited from February 2012 to July 2013, underwent 2 passes with a standard 25G needle for cytologic analysis, and were randomized, 30 per group, to undergo 2 passes with 22Gpc (1 pass each for cytology and histology), using SST or CST.
Groups:
- Standard Suction Technique (SST): P30 participants randomized to SST (Standard Suction Technique)
- Capillary Suction Technique (CST): 30 participants randomized to CST (Capillary Suction Technique
Period: Overall Study
Arm/Group | Standard Suction Technique (SST) | Capillary Suction Technique (CST)
Started | 30 | 30
2 Passes With 25G for Cytology | 30 | 30
1 Pass With 22Gpc for Cytology | 29 (1 participant's pass could not be performed) | 30
1 Pass With 22Gpc for Histology | 27 (3 participants passes could not be performed) | 29 (1 participant's pass could not be performed)
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Suction Technique (SST): SST: 2 passes with 25G for cytology, 1 pass each with 22Gpc for cytology and histology. Diagnostic adequacy scores compared by technique and by needle
- Capillary Suction Technique (CST): CST: 2 passes with 25G for cytology, 1 pass each with 22Gpc for cytology and histology. Diagnostic adequacy scores compared by technique and by needle
- Total: Total of all reporting groups
Arm/Group | Standard Suction Technique (SST) | Capillary Suction Technique (CST) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 19 | 31
  >=65 years | 18 | 11 | 29
Age, Continuous [Mean (Full Range); unit: years] | 65 [31 to 78] | 61 [24 to 85] | 63 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 16 | 19 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 26 | 22 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Diagnostic Adequacy Scores With SST vs. CST for Cytologic Diagnosis Using a 22G Core Needle.
Description: The main outcome measure of the study was the diagnostic adequacy of the 22Gpc using SST and CST. The cytologic diagnostic adequacy of 22Gpc was also compared to the standard 25 G needle. Each participant underwent 4 study passes, 2 passes with a standard 25 G needle using SST, plus a random assignment to one of two groups for 2 passes with the 22Gpc (1 pass for cytologic and 1 pass for histologic analysis) using SST (group 1) or CST (group 2). Diagnostic adequacy was defined as the ability to procure cytological aspirates or histological core tissue samples that were sufficient for diagnostic interpretation.
Time Frame: Each EGD EUS-FNA endoscopy procedure takes about 1 hour. Each needle pass takes about 1-2 minutes.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Suction Technique (SST) Cytology: 1 pass with 22Gpc for cytology, 1 pass with 22Gpc for histology using SST or CST. Diagnostic adequacy scores compared by technique for cytology and histology.
- Capillary Suction Technique (CST): 30 participants randomized to CST (Capillary Suction Technique)
Arm/Group | Standard Suction Technique (SST) Cytology | Capillary Suction Technique (CST)
Number analyzed (Participants) | 29 | 30
Participants
  All pancreas masses: Score 0 or 1 | 5 | 6
  All pancreas masses: Score 2 or 3 | 24 | 24
  All pancreas masses: Score 3 | 23 | 21
  Adenocarcinoma: Score 0 or 1 | 4 | 5
  Adenocarcinoma: Score 2 or 3 | 18 | 18
  Adenocarcinoma: Score 3 | 17 | 17

2. Primary Outcome: Comparison of Diagnostic Adequacy Scores With SST vs. CST for Histologic Diagnosis Using a 22G Core Needle.
Description: The main outcome measure of the study was the diagnostic adequacy of the 22Gpc using SST versus CST on EUS-FNA. The cytologic diagnostic adequacy of 22Gpc was also compared to the standard 25G needle. Diagnostic adequacy was defined as the ability to procure cytological aspirates or histological core tissue samples that were sufficient for diagnostic interpretation. Two cytopathologists, blinded to needle type and technique, reviewed and graded all the study slides. Cytologic diagnostic adequacy of each pass was graded on a semiquantitative scale from 0 to 3 based on sample cellularity. A score of 2 (estimated cell count > 500 cells) or 3 (estimated cell count > 1000 cells) was considered adequate for diagnosis; a score of 3 was most desirable. A score < 2 was considered inadequate. Histologic diagnostic adequacy was graded as either an adequate (score 2 or 3) or inadequate specimen for diagnosis.
Time Frame: Each EGD EUS-FNA endoscopy procedure takes about 1 hour. Each needle pass takes about 1-2 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Standard Suction Technique (SST) Histology: 1 pass with 22Gpc for histology using SST. Diagnostic adequacy scores compared by technique for histology.
- Capillary Suction Technique (CST) Histology: 1 pass with 22Gpc for histology using CST. Diagnostic adequacy scores compared by technique for histology.
Arm/Group | Standard Suction Technique (SST) Histology | Capillary Suction Technique (CST) Histology
Number analyzed (Participants) | 27 | 29
Participants
  All pancreas masses: Score 0 or 1 | 8 | 9
  All pancreas masses: Score 2 or 3 | 19 | 20
  Adenocarcinoma: Score 0 or 1 | 5 | 8
  Adenocarcinoma: Score 2 or 3 | 15 | 14

3. Secondary Outcome: Comparison of Diagnostic Adequacy of Single Pass With 22G Core Needle and Standard 25G Needle for Cytologic Diagnosis
Description: The cytologic diagnostic adequacy of 22Gpc was compared to the standard 25G needle. Diagnostic adequacy was defined as the ability to procure cytological aspirates that were sufficient for diagnostic interpretation. Two cytopathologists, blinded to needle type and technique, reviewed and graded all the study slides. Cytologic diagnostic adequacy of each pass was graded on a semiquantitative scale from 0 to 3 based on sample cellularity. A score of 2 (estimated cell count > 500 cells) or 3 (estimated cell count > 1000 cells) was considered adequate for diagnosis; a score of 3 was most desirable. A score < 2 was considered inadequate.
Time Frame: Each EGD EUS-FNA endoscopy procedure takes about 1 hour. Each needle pass takes about 1-2 minutes
Measure: Count of Participants; unit: Participants
Groups:
- 22G Procore Needle; Standard 25G Needle: All patients: comparison of diagnostic adequacy of a single pass with a 22Gpc needle versus best of 2 passes with a standard 25G needle for cytological diagnosis.
Arm/Group | 22G Procore Needle | Standard 25G Needle
Number analyzed (Participants) | 59 | 60
Participants
  All pancreas masses: Score 2 or 3 | 48 | 57
  All pancreas masses: Score 3 | 44 | 45
  Adenocarcinoma: Score 2 or 3 | 36 | 43
  Adenocarcinoma: Score 3 | 34 | 34

ADVERSE EVENTS:
Time Frame: Electronic chart review was performed by the PI for any adverse events recorded within 2 weeks of the procedure
Groups:
- Standard Suction Technique (SST); Capillary Suction Technique (CST): Participants who are referred for EUS-FNA and consented will have their examination performed using two different needles: with the standard 22-gauge or 25-gauge straight hollow core needle
Arm/Group | Standard Suction Technique (SST) | Capillary Suction Technique (CST)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT01598194/Prot_SAP_000.pdf